CLINICAL TRIAL: NCT04220697
Title: Behavioural and Neurophysiological Measurements for the Assessment of Central Sensitisation and Postoperative Pain
Brief Title: Central Sensitisation and Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: POSTOP pain
Record Dates: First submitted 2020-01-06; First posted 2020-01-07 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Thoracotomy; Hyperalgesia; Hyperalgesia, Secondary; Central Sensitisation; Electroencephalography; Persistent Postsurgical Pain; Humans
MeSH Terms: conditions — Hyperalgesia; Pain, Postoperative | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergo lateral thoracotomy for primary lung cancer (Experimental): 1. Electroencephalography (EEG) will be acquired before surgery
  2. Questionnaires assessing psychological status of the patients before and after surgery
  3. High frequency electrical stimulation of the skin (HFS) will be delivered before surgery
  4. Quantification of mechanical sensitivity after HFS and after surgery
  Interventions: Other: electroencephalography (EEG); Other: questionnaires; Other: high frequency electrical stimulation of the forearm skin (HFS); Other: cutaneous mechanical pinprick stimulation

INTERVENTIONS:
Other: electroencephalography (EEG) — recording of resting state EEG using 64 surface electrodes
Other: questionnaires — Hospital Anxiety Depression Scale (HADS) Neuropathic Pain questionnaire (DN4) Brief Pain Inventory (BPI) Fatigue Assessment Scale (FAS)
Other: high frequency electrical stimulation of the forearm skin (HFS) — HFS consists of transcutaneous electrical stimuli delivered as 42 Hz trains (pulse width: 2 ms) lasting 1 s. The trains are repeated 12 times. Each train is separated by 10 seconds.
Other: cutaneous mechanical pinprick stimulation — Mechanical pinprick stimuli will be applied manually by the operator on the skin using a mechanical stimulator (maximum weight 128 mN).

SUMMARY:
One out of 10 patients undergoing surgery develops persistent post-surgical pain (PPSP). Unfortunately, available therapies for treating this pain have limited success. It is therefore of great importance to find strategies to prevent PPSP. The goal of this project is to find new screening tools that identify patients that are at risk for developing PPSP.

Tissue injury and inflammation following surgery increase the excitability of spinal nociceptive neurons ("central sensitisation", CS) with pain hypersensitivity as consequence. It is thought that CS plays an important role in persistent pain.

The first objective of this project is to assess in human patients if the propensity to develop CS manifested as secondary hyperalgesia before surgery is predictive for PPSP.

In addition, we will test if the frequency content of the resting-state EEG reflecting the initial state of the brain will be related to the propensity for developing CS and to the presence of PPSP at two months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a lateral thoracotomy as treatment for primary lung cancer
* Ability to provide written informed consent

Exclusion Criteria:

* Evidence for a clinically-significant alteration of the skin of the volar forearms
* Pregnancy
* Having a pacemaker or implanted cardiac defibrillator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
mechanical pinprick perceived intensity | 1 day before surgery
  magnitude of the increase in sensitivity to mechanical pinprick stimuli after HFS
area of increased mechanical pinprick sensitivity | 1 day before surgery
  spatial extent of the increased sensitivity to mechanical pinprick stimuli after HFS
resting state EEG | 1 week before surgery
  frequency content of the resting state EEG

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Lacroix, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (2):
- Belgium (2):
  - Department of Surgery, Brussels
  - Saint Luc Hospital, Brussels

IPD SHARING:
Plan to Share IPD: No